CLINICAL TRIAL: NCT04409288
Title: Patient Preference of Apalutamide Versus Enzalutamide in Patients With Recurrent or Metastatic Hormone-Sensitive Prostate Cancer: An Open-label, Randomized, Cross-Over Trial.
Brief Title: Patient Preference of Apalutamide Versus Enzalutamide in Patients With Recurrent or Metastatic Hormone-Sensitive Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Endpoint reached
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 56021927PCR3012
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: Patient Preference
MeSH Terms: conditions — Prostatic Neoplasms; Patient Preference | interventions — apalutamide; enzalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): Apalutamide followed by Enzalutamide Study participants will receive 12 weeks of oral apalutamide (240mg) daily, followed by five weeks of washout period, and then 12 weeks of oral enzalutamide (160mg) daily.
  Interventions: Drug: Apalutamide; Drug: Enzalutamide
- Group B (Experimental): Enzalutamide followed by Apalutamide Study participants will receive 12 weeks of oral enzalutamide (160mg) daily, followed by five weeks of washout period, and then 12 weeks of oral apalutamide (240mg) daily.
  Interventions: Drug: Apalutamide; Drug: Enzalutamide

INTERVENTIONS:
Drug: Apalutamide — Androgen receptor inhibitor.
Drug: Enzalutamide — Androgern receptor inhibitor

SUMMARY:
This is a prospective, open-label, randomized, controlled, cross-over trial assessing patient preference for apalutamide versus enzalutamide in 146 male patients with recurrent or metastatic hormone-sensitive prostate cancer. The primary objective is to investigate whether there is any difference in patient preference between apalutamide and enzalutamide in patients with recurrent or metastatic hormone-sensitive prostate cancer.

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized, controlled, cross-over trial assessing patient preference for apalutamide versus enzalutamide in 146 male patients with recurrent or metastatic hormone-sensitive prostate cancer The primary outcome is patient preference, which serves as an indicator covering different aspects of treatment-related effects, and this would be most important in a patient's perspective. The quality of life, psychological and cognitive changes following apalutamide and enzalutamide in a comprehensive manner will be investigated.

Patient will receive two 12-weeks treatment periods with a 5-week wash-out period between the treatment periods. Patients will receive Apalutamide and Enzulutamide sequentially. Patient, physician and caregiver preferences will be assessed at the end of the second treatment period. Other secondary outcomes on health-related quality of life measures, psychological assessment scores and cognitive assessment scores shall be assessed before and the end of first treatment and second treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or above with informed consent
2. Histological diagnosis of adenocarcinoma of the prostate without neuroendocrine differentiation, signet cell, or small cell features
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
4. Androgen deprivation therapy started at least 28 days prior to randomization
5. Patients should be having one of the following diseases and treatment conditions:

   1. Recurrent prostate cancer following radical prostatectomy or radiotherapy, which do not fall into high-risk or high-volume categories
   2. Metastatic hormone-sensitive prostate cancer, which do not fall into high-risk or high-volume categories

Exclusion Criteria:

1. Patients with high-volume metastatic hormone-sensitive prostate cancer, defined by the presence of visceral metastases or four or more bone lesions with at least one beyond the vertebral bodies and pelvis
2. Patients with high-risk metastatic hormone-sensitive prostate cancer, defined by having at least two of the three following factors - a Gleason score above 7, having at least 3 bone metastasis or presence of measurable visceral metastasis
3. Presence of brain metastasis
4. Use of bisphosphonate or denosumab within 28 days prior to randomization
5. Use of older anti-androgens, including flutamide and bicalutamide, for flare protection, within 28 days prior to randomization
6. Prior use of chemotherapy, immunotherapy, radiopharmaceutical agents, CYP17 inhibitors (e.g. abiraterone acetate), enzalutamide or apalutamide for the treatment of prostate cancer or prior participation in a clinical trial of an investigational agent that inhibits the androgen receptor or androgen synthesis
7. History of seizure or any condition that may predispose to seizure (e.g., neurological disorder, prior cortical stroke or significant brain trauma)
8. Use of an investigational agent within 4 weeks of randomization
9. Hypersensitivity reaction to the active pharmaceutical ingredient
10. Clinically significant cardiovascular disease including the following:

    1. Myocardial infarction within 6 months before screening;
    2. Uncontrolled angina within 3 months before screening;
    3. Congestive heart failure New York Heart Association class 3 or 4, or a history of congestive heart failure New York Heart Association class 3 or 4, unless a screening echocardiogram or multigated acquisition scan performed within 3 months before randomization demonstrates a left ventricular ejection fraction ≥ 50%;
    4. History of clinically significant ventricular arrhythmias (e.g. sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes);
    5. History of Mobitz II second-degree or third-degree heart block without a permanent pacemaker in place;
    6. Hypotension as indicated by systolic blood pressure < 86 millimeters of mercury (mm Hg) at screening;
    7. Bradycardia as indicated by a heart rate of < 45 beats per minute on the screening electrocardiogram and on physical examination;
    8. Uncontrolled hypertension as indicated by systolic blood pressure > 170 mm Hg or diastolic blood pressure > 105 mm Hg at screening
11. Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer disease within 3 months before randomization)
12. Major surgery within 28 days of randomization
13. Any concurrent disease, infection, or comorbid condition that interferes with the ability of the patient to participate in the trial, which places the patient at undue risk, or complicates the interpretation of data, in the opinion of the investigator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 74 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Patient Preference Questionnaire | Week 29 (at the end of second treatment)
  This Patient Preference Questionnaire consists of 4 questions, assessing the patients preference on Apalutamide verse Enzalutamide, the factors that had an influence on their treatment preference, the most important reason for their preference and the side effect of first treatment and second treatment.

SECONDARY OUTCOMES:
The side effect profile as assessed Patient Preference Questionnaire | Baseline to week 29 (the end of the study)
  In Patient Preference Questionnaire, participants completed a sideffect checklist.
Physician Preference Questionnaire | Week 29 (at the end of second treatment)
  This Physician Preference Questionnaire consists of 3 questions, assessing the physicians preference on Apalutamide verse Enzalutamide, the factors that had an influence on their treatment preference, the most important reason for their preference.
Caregiver Preference Questionnaire | Week 29 (at the end of second treatment)
  This Caregiver Preference Questionnaire consists of 3 questions, assessing the caregivers preference on Apalutamide verse Enzalutamide, the factors that had an influence on their treatment preference, the most important reason for their preference.
The Functional Assessment of Cancer Therapy-Prostate Questionnaire (FACT-P) | Week 0 (before start of first treatment period), Week 12 (end of first treatment period), week 17 (before start of second treatment period) and Week 29 (end of second treatment period).
  This is a 39-item questionnaire assessing five domains including Physical Well-Being, Social and Family Well-Being, Emotional Well-Being, Functional Well-Being and Prostate Cancer Subscale.The higher the score, the better the QOL
Quality of life measured by EurolQol instrument (EQ-5D-5L) | Week 0 (before start of first treatment period), Week 12 (end of first treatment period), week 17 (before start of second treatment period) and Week 29 (end of second treatment period
  This questionnaire consists of two parts, namely the EQ-5D-5L Descriptive System and the EQ Visual Analog Scale, the higher the score the better in quality of life
FACT-Cognitive Function Version 3 (FACT-Cog) | Week 0 (before start of first treatment period), Week 12 (end of first treatment period), week 17 (before start of second treatment period) and Week 29 (end of second treatment period
  This is a well-established 37-item questionnaire assessing patients' perceived cognitive impairments, perceived cognitive abilities, noticeability or comments from others, and impact of cognitive changes on quality of life. The higher the score, the better the QOL.
Brief Fatigue Inventory (BFI) | Week 0 (before start of first treatment period), Week 12 (end of first treatment period), week 17 (before start of second treatment period) and Week 29 (end of second treatment period
  This is a well-established 9-item questionnaire assessing patients' degree of fatigue.The higher the score, the higher fatigue level

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huggins C, Hodges CV. Studies on prostatic cancer. I. The effect of castration, of estrogen and androgen injection on serum phosphatases in metastatic carcinoma of the prostate. CA Cancer J Clin. 1972 Jul-Aug;22(4):232-40. doi: 10.3322/canjclin.22.4.232. No abstract available. PMID 4625049
- [Background] Walsh PC. Immediate versus deferred treatment for advanced prostatic cancer: initial results of the Medical Research Council trial. The Medical Research Council Prostate Cancer Working Party Investigators Group. J Urol. 1997 Oct;158(4):1623-4. No abstract available. PMID 9302187
- [Background] Ryan CJ, Smith MR, de Bono JS, Molina A, Logothetis CJ, de Souza P, Fizazi K, Mainwaring P, Piulats JM, Ng S, Carles J, Mulders PF, Basch E, Small EJ, Saad F, Schrijvers D, Van Poppel H, Mukherjee SD, Suttmann H, Gerritsen WR, Flaig TW, George DJ, Yu EY, Efstathiou E, Pantuck A, Winquist E, Higano CS, Taplin ME, Park Y, Kheoh T, Griffin T, Scher HI, Rathkopf DE; COU-AA-302 Investigators. Abiraterone in metastatic prostate cancer without previous chemotherapy. N Engl J Med. 2013 Jan 10;368(2):138-48. doi: 10.1056/NEJMoa1209096. Epub 2012 Dec 10. PMID 23228172
- [Background] Fizazi K, Scher HI, Molina A, Logothetis CJ, Chi KN, Jones RJ, Staffurth JN, North S, Vogelzang NJ, Saad F, Mainwaring P, Harland S, Goodman OB Jr, Sternberg CN, Li JH, Kheoh T, Haqq CM, de Bono JS; COU-AA-301 Investigators. Abiraterone acetate for treatment of metastatic castration-resistant prostate cancer: final overall survival analysis of the COU-AA-301 randomised, double-blind, placebo-controlled phase 3 study. Lancet Oncol. 2012 Oct;13(10):983-92. doi: 10.1016/S1470-2045(12)70379-0. Epub 2012 Sep 18. PMID 22995653
- [Background] Scher HI, Fizazi K, Saad F, Taplin ME, Sternberg CN, Miller K, de Wit R, Mulders P, Chi KN, Shore ND, Armstrong AJ, Flaig TW, Flechon A, Mainwaring P, Fleming M, Hainsworth JD, Hirmand M, Selby B, Seely L, de Bono JS; AFFIRM Investigators. Increased survival with enzalutamide in prostate cancer after chemotherapy. N Engl J Med. 2012 Sep 27;367(13):1187-97. doi: 10.1056/NEJMoa1207506. Epub 2012 Aug 15. PMID 22894553
- [Background] Beer TM, Armstrong AJ, Rathkopf DE, Loriot Y, Sternberg CN, Higano CS, Iversen P, Bhattacharya S, Carles J, Chowdhury S, Davis ID, de Bono JS, Evans CP, Fizazi K, Joshua AM, Kim CS, Kimura G, Mainwaring P, Mansbach H, Miller K, Noonberg SB, Perabo F, Phung D, Saad F, Scher HI, Taplin ME, Venner PM, Tombal B; PREVAIL Investigators. Enzalutamide in metastatic prostate cancer before chemotherapy. N Engl J Med. 2014 Jul 31;371(5):424-33. doi: 10.1056/NEJMoa1405095. Epub 2014 Jun 1. PMID 24881730
- [Background] Parker C, Nilsson S, Heinrich D, Helle SI, O'Sullivan JM, Fossa SD, Chodacki A, Wiechno P, Logue J, Seke M, Widmark A, Johannessen DC, Hoskin P, Bottomley D, James ND, Solberg A, Syndikus I, Kliment J, Wedel S, Boehmer S, Dall'Oglio M, Franzen L, Coleman R, Vogelzang NJ, O'Bryan-Tear CG, Staudacher K, Garcia-Vargas J, Shan M, Bruland OS, Sartor O; ALSYMPCA Investigators. Alpha emitter radium-223 and survival in metastatic prostate cancer. N Engl J Med. 2013 Jul 18;369(3):213-23. doi: 10.1056/NEJMoa1213755. PMID 23863050
- [Background] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- [Background] Sweeney CJ, Chen YH, Carducci M, Liu G, Jarrard DF, Eisenberger M, Wong YN, Hahn N, Kohli M, Cooney MM, Dreicer R, Vogelzang NJ, Picus J, Shevrin D, Hussain M, Garcia JA, DiPaola RS. Chemohormonal Therapy in Metastatic Hormone-Sensitive Prostate Cancer. N Engl J Med. 2015 Aug 20;373(8):737-46. doi: 10.1056/NEJMoa1503747. Epub 2015 Aug 5. PMID 26244877
- [Background] James ND, Sydes MR, Clarke NW, Mason MD, Dearnaley DP, Spears MR, Ritchie AW, Parker CC, Russell JM, Attard G, de Bono J, Cross W, Jones RJ, Thalmann G, Amos C, Matheson D, Millman R, Alzouebi M, Beesley S, Birtle AJ, Brock S, Cathomas R, Chakraborti P, Chowdhury S, Cook A, Elliott T, Gale J, Gibbs S, Graham JD, Hetherington J, Hughes R, Laing R, McKinna F, McLaren DB, O'Sullivan JM, Parikh O, Peedell C, Protheroe A, Robinson AJ, Srihari N, Srinivasan R, Staffurth J, Sundar S, Tolan S, Tsang D, Wagstaff J, Parmar MK; STAMPEDE investigators. Addition of docetaxel, zoledronic acid, or both to first-line long-term hormone therapy in prostate cancer (STAMPEDE): survival results from an adaptive, multiarm, multistage, platform randomised controlled trial. Lancet. 2016 Mar 19;387(10024):1163-77. doi: 10.1016/S0140-6736(15)01037-5. Epub 2015 Dec 21. PMID 26719232
- [Background] Clegg NJ, Wongvipat J, Joseph JD, Tran C, Ouk S, Dilhas A, Chen Y, Grillot K, Bischoff ED, Cai L, Aparicio A, Dorow S, Arora V, Shao G, Qian J, Zhao H, Yang G, Cao C, Sensintaffar J, Wasielewska T, Herbert MR, Bonnefous C, Darimont B, Scher HI, Smith-Jones P, Klang M, Smith ND, De Stanchina E, Wu N, Ouerfelli O, Rix PJ, Heyman RA, Jung ME, Sawyers CL, Hager JH. ARN-509: a novel antiandrogen for prostate cancer treatment. Cancer Res. 2012 Mar 15;72(6):1494-503. doi: 10.1158/0008-5472.CAN-11-3948. Epub 2012 Jan 20. PMID 22266222
- [Background] Smith MR, Saad F, Chowdhury S, Oudard S, Hadaschik BA, Graff JN, Olmos D, Mainwaring PN, Lee JY, Uemura H, Lopez-Gitlitz A, Trudel GC, Espina BM, Shu Y, Park YC, Rackoff WR, Yu MK, Small EJ; SPARTAN Investigators. Apalutamide Treatment and Metastasis-free Survival in Prostate Cancer. N Engl J Med. 2018 Apr 12;378(15):1408-1418. doi: 10.1056/NEJMoa1715546. Epub 2018 Feb 8. PMID 29420164
- [Background] Esper P, Mo F, Chodak G, Sinner M, Cella D, Pienta KJ. Measuring quality of life in men with prostate cancer using the functional assessment of cancer therapy-prostate instrument. Urology. 1997 Dec;50(6):920-8. doi: 10.1016/S0090-4295(97)00459-7. PMID 9426724
- [Background] Rathkopf DE, Morris MJ, Fox JJ, Danila DC, Slovin SF, Hager JH, Rix PJ, Chow Maneval E, Chen I, Gonen M, Fleisher M, Larson SM, Sawyers CL, Scher HI. Phase I study of ARN-509, a novel antiandrogen, in the treatment of castration-resistant prostate cancer. J Clin Oncol. 2013 Oct 1;31(28):3525-30. doi: 10.1200/JCO.2013.50.1684. Epub 2013 Sep 3. PMID 24002508
- [Background] Wong CK, Choi EP, Tsu JH, Ho BS, Ng AT, Chin WY, Yiu MK. Psychometric properties of Functional Assessment of Cancer Therapy-Prostate (FACT-P) in Chinese patients with prostate cancer. Qual Life Res. 2015 Oct;24(10):2397-402. doi: 10.1007/s11136-015-0993-8. Epub 2015 Apr 16. PMID 25877953
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Janssen MF, Pickard AS, Golicki D, Gudex C, Niewada M, Scalone L, Swinburn P, Busschbach J. Measurement properties of the EQ-5D-5L compared to the EQ-5D-3L across eight patient groups: a multi-country study. Qual Life Res. 2013 Sep;22(7):1717-27. doi: 10.1007/s11136-012-0322-4. Epub 2012 Nov 25. PMID 23184421
- [Background] Costa DSJ, Loh V, Birney DP, Dhillon HM, Fardell JE, Gessler D, Vardy JL. The Structure of the FACT-Cog v3 in Cancer Patients, Students, and Older Adults. J Pain Symptom Manage. 2018 Apr;55(4):1173-1178. doi: 10.1016/j.jpainsymman.2017.12.486. Epub 2017 Dec 30. PMID 29291932
- [Background] Mendoza TR, Wang XS, Cleeland CS, Morrissey M, Johnson BA, Wendt JK, Huber SL. The rapid assessment of fatigue severity in cancer patients: use of the Brief Fatigue Inventory. Cancer. 1999 Mar 1;85(5):1186-96. doi: 10.1002/(sici)1097-0142(19990301)85:53.0.co;2-n. PMID 10091805
- [Background] Escudier B, Porta C, Bono P, Powles T, Eisen T, Sternberg CN, Gschwend JE, De Giorgi U, Parikh O, Hawkins R, Sevin E, Negrier S, Khan S, Diaz J, Redhu S, Mehmud F, Cella D. Randomized, controlled, double-blind, cross-over trial assessing treatment preference for pazopanib versus sunitinib in patients with metastatic renal cell carcinoma: PISCES Study. J Clin Oncol. 2014 May 10;32(14):1412-8. doi: 10.1200/JCO.2013.50.8267. Epub 2014 Mar 31. PMID 24687826
- [Background] Senn S, Stevens L, Chaturvedi N. Repeated measures in clinical trials: simple strategies for analysis using summary measures. Stat Med. 2000 Mar 30;19(6):861-77. doi: 10.1002/(sici)1097-0258(20000330)19:63.0.co;2-f. PMID 10734289